CLINICAL TRIAL: NCT01277458
Title: Accuracy of Ethnicity Recording in MSM Patients With HIV of Non-White Ethnicity in London
Brief Title: Ethnicity Data in HIV Positive Men Who Have Sex With Men
Status: Withdrawn | Type: Observational
Why Stopped: Unable to recruit participants
Sponsor: Public Health England (Other Government)
Responsible Party: Sponsor
Other Study IDs: EthMSM01
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2010-12

CONDITIONS: HIV
Keywords: HIV; MSM; Ethnicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non white HIV positive men who have sex with men

SUMMARY:
Are there differences between the way that non-White men who have sex with men living in London with HIV describe their own ethnicity and the way in which their ethnic group is recorded in NHS clinics? We aim to describe the way in which clinics in London currently record a patient's ethnic group. Without accurate data for an individual's ethnic group we are unable to draw meaningful conclusions about their experiences of HIV care. It may be the case that patients from particular ethnic groups require specific ways of monitoring and treating their HIV but without knowing if these people are in a particular group any services directed to them may be wasted or underused.

DETAILED DESCRIPTION:
HIV Doctors will be identified at each of the London HIV treatment centres and details of the project will be communicated to them via email.

These doctors will then be sent paper copies of the patient information sheets (PIS), patient questionnaires and clinician questionnaires.

Eligible patients (i.e. men having sex with men with HIV from non-white ethnic groups) will be identified by their doctors and will be asked to read the PIS and complete the questionnaire. This will be a single questionnaire and no follow up for the patient will be required. No personal information (e.g. date of birth, hospital number) will be recorded. Eligible patients will be all those coming to clinic for HIV care between 1st June and 31st of July 2011. Based on estimates from 2009 data held by the HPA, each doctor will on average be asked to recruit 30 patients over the two month period.

The questionnaire will ask questions regarding self description of ethnicity, sexuality, parents' ethnicity, country of birth and other countries of residency (if relevant). It is anticipated that to read the PIS and complete the questionnaire should take no longer than 15 minutes.

The doctor will then return the paper questionnaire (in an addressed envelope supplied) to Dr Williams. Dr Williams will then bring together and analyse the data from the questionnaires and write up her findings for publication and presentation at a national conference.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with HIV
* Male patients who have ever had sex with other men (bi- or homosexual to both be included)
* Patients of non-white ethnicity (patients described as being of "mixed" or "other" ethnicity are to be included)

Exclusion Criteria:

* Female patients
* Male patients who have only ever had sex with women
* Patients whose ethnicity is described as "White"
* Patients unable to read or understand the written questionnaire

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 400 Non-White HIV positive Men who have sex with men
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-03 (Estimated); Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of misclassification of ethnicity for non-White MSM with HIV living in London | end of study (2 months)

SECONDARY OUTCOMES:
• Prevalence of individual non-White self-identified ethnicity groups in MSM with HIV in London | End of study (2 months)
Description of current clinic practice for ethnicity data recording | End of study (2 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom